CLINICAL TRIAL: NCT00118755
Title: A Randomized, Open-label Study of the Effect of 2 Different Treatment Schedules of Xeloda With Eloxatin and Avastin on Progression-free Survival in Treatment-naïve Patients With Locally Advanced or Metastatic Colorectal Cancer
Brief Title: A Study of Two Different Schedules of Xeloda (Capecitabine) as First Line Therapy in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Disclosures Group, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18491
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Results first posted 2011-03-03 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Bevacizumab

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: capecitabine; Drug: Oxaliplatin; Drug: bevacizumab
- 2 (Active Comparator)
  Interventions: Drug: capecitabine; Drug: Oxaliplatin; Drug: bevacizumab

INTERVENTIONS:
Drug: capecitabine — 850 mg/m^2 po bid on Days 1-14 of each 3-week cycle
  Arms: 1
Drug: Oxaliplatin — 130 mg/m^2 IV on Day 1 of each 3-week cycle
  Arms: 1
Drug: bevacizumab — 7.5 mg/kg IV on Day 1 of each 3-week cycle
  Arms: 1
Drug: capecitabine — 1500 mg/m^2 po bid on Days 1-7 of each 2-week cycle
  Arms: 2
Drug: Oxaliplatin — 85 mg/m^2 IV on Day 1 of each 2-week cycle
  Arms: 2
Drug: bevacizumab — 5 mg/kg IV on Day 1 of each 2-week cycle
  Arms: 2

SUMMARY:
This 2-arm study evaluated the efficacy and safety of 2 different treatment schedules of oral Xeloda with intravenous (IV) Eloxatin (oxaliplatin) and IV bevacizumab (Avastin) as a first-line treatment in patients with locally advanced or metastatic colorectal cancer. Patients were randomized to receive either: 1) Xeloda 850 mg/m^2 orally twice a day (po bid) on Days 1-14, oxaliplatin 130 mg/m^2 IV on Day 1, and Avastin 7.5 mg/kg IV on Day 1 of each 3-week cycle; or 2) Xeloda 1500 mg/m^2 po bid on Days 1-7, oxaliplatin 85 mg/m^2 IV on Day 1 and Avastin 5 mg/kg IV on Day 1 of each 2-week cycle. The anticipated time on study treatment was 1-2 years, and the target sample size was 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or inoperable locally advanced colorectal cancer
* >=1 measurable target lesion

Exclusion Criteria:

* Previous systemic therapy for advanced or metastatic disease
* Previous treatment with bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2005-07; Primary Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

RESULTS

PARTICIPANT FLOW:
Groups:
- XELOX Q3W + Bevacizumab: Capecitabine 850 mg/m^2 twice-daily was given orally. Bevacizumab 7.5 mg/kg via 30-90 minute intravenous (IV) infusion was administered on day 1 every three weeks prior to administration of oxaliplatin.
  Oxaliplatin 130 mg/m^2 via 2-hour IV infusion was administered on day 1 every 3 weeks.
- XELOX Q2W + Bevacizumab: Capecitabine 1500 mg/m^2 twice-daily was given orally. Bevacizumab 5 mg/kg via 30-90 minute intravenous (IV) infusion was administered on day 1 every two weeks prior to administration of oxaliplatin.
  Oxaliplatin 85 mg/m^2 via 2-hour IV infusion was administered on day 1 every 2 weeks.
Period: Overall Study
Arm/Group | XELOX Q3W + Bevacizumab | XELOX Q2W + Bevacizumab
Started | 217 | 218
Safety Population | 208 | 211
Completed | 7 | 3
Not Completed | 210 | 215

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XELOX Q3W + Bevacizumab | XELOX Q2W + Bevacizumab | Total
Number analyzed (Participants) | 217 | 218 | 435
Age Continuous [Mean (Standard Deviation); unit: years] | 60.6 (11.45) | 60.8 (12.17) | 60.7 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 96 | 185
  Male | 128 | 122 | 250

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was defined as the time from the date of randomization to the first occurrence of having documented disease progression or death due to any cause, whichever comes first. Progression was based on tumor assessments made by the investigators according to Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: Time to disease progression or death (through follow-up phase)
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | XELOX Q3W + Bevacizumab | XELOX Q2W + Bevacizumab
Number analyzed (Participants) | 217 | 218
Days | 287 [234 to 329] | 273 [231 to 313]
Statistical Analysis 1: Comparison: XELOX Q3W + Bevacizumab vs XELOX Q2W + Bevacizumab; Test type: Superiority or Other; p = 0.3883, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.67 to 1.17]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of randomization to the date of death, for any cause.
Time Frame: Time to death (through follow-up phase): Approximate Median of 718 days
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | XELOX Q3W + Bevacizumab | XELOX Q2W + Bevacizumab
Number analyzed (Participants) | 217 | 218
Days | 852 [605 to 1052] | 662 [595 to 762]
Statistical Analysis 1: Comparison: XELOX Q3W + Bevacizumab vs XELOX Q2W + Bevacizumab; Test type: Superiority or Other; p = 0.2458, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.64 to 1.12]

3. Secondary Outcome: Best Overall Clinical Response
Description: Overall response rate was assessed according to RECIST (the best response recorded from the time of randomization to the first CR or PR. The patient's overall best response was complete response (CR), partial response (PR) (CR and PR considered "responders"), stable disease (SD), or progressive disease (PD). To be assigned a status of complete response (CR) or partial response (PR), changes in tumor measurements were confirmed by repeat assessments performed no less than 4 weeks after the criteria for response were first met.
Time Frame: Through follow-up phase: Approximate Median of 318 days
Population: Intent-to-treat population
Measure: Number; unit: Patients
Arm/Group | XELOX Q3W + Bevacizumab | XELOX Q2W + Bevacizumab
Number analyzed (Participants) | 217 | 218
Patients
  Nonresponders (without CR or PR) | 145 | 167
  Responders (with CR or PR) | 72 | 51
  Complete Response (CR) | 2 | 3
  Partial Response (PR) | 70 | 48
Statistical Analysis 1: Comparison: XELOX Q3W + Bevacizumab vs XELOX Q2W + Bevacizumab; Test type: Superiority or Other; Difference in Response Rate = 9.8, 95% CI [0.9 to 18.7] — 95% Wald asymptotic CI using normal approximation (continuity corrected)

4. Secondary Outcome: Duration of Overall Clinical Response (CR or PR)
Description: Among tumor responders (i.e., patients with overall best response of CR or PR), duration of overall response was measured from the time criteria were first met for CR or PR (whichever status was recorded first) to the date of either recurrent/progressive disease was objectively documented or death from any cause.
Time Frame: Time to Disease Progression or Death (through follow-up phase): Approximate Median of 302 days
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Days to event
Arm/Group | XELOX Q3W + Bevacizumab | XELOX Q2W + Bevacizumab
Number analyzed (Participants) | 217 | 218
Days to event | 281 [225 to 397] | 316 [244 to 522]
Statistical Analysis 1: Comparison: XELOX Q3W + Bevacizumab vs XELOX Q2W + Bevacizumab; Test type: Superiority or Other; p = 0.6294, Log Rank; Hazard Ratio (HR) = 1.14, 95% CI [0.66 to 1.97]

ADVERSE EVENTS:
Description: Safety Population = Received at least 1 dose of study medication. XELOX Q3W + Bevacizumab n=208 XELOX Q2W + Bevacizumab n=211
Arm/Group | XELOX Q3W + Bevacizumab | XELOX Q2W + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 84/208 | 94/211
Other Adverse Events (participants affected / at risk) | 202/208 | 206/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XELOX Q3W + Bevacizumab (N=208) | XELOX Q2W + Bevacizumab (N=211)
Diarrhoea (Gastrointestinal disorders) | 20 | 22
Abdominal Pain (Gastrointestinal disorders) | 3 | 6
Small Intestinal Obstruction (Gastrointestinal disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 4 | 4
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 3 | 3
Ileus (Gastrointestinal disorders) | 1 | 3
Colitis (Gastrointestinal disorders) | 2 | 1
Enteritis (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Rectal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Caecitis (Gastrointestinal disorders) | 1 | 0
Colonic Obstruction (Gastrointestinal disorders) | 0 | 1
Colonic Pseudo-Obstruction (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Ileitis (Gastrointestinal disorders) | 1 | 0
Ileus Paralytic (Gastrointestinal disorders) | 0 | 1
Inflammatory Bowel Disease (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0
Mechanical Ileus (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Pancreatitus (Gastrointestinal disorders) | 0 | 1
Pancreatitus Acute (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Small Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 21 | 18
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Gastrointestinal disorders) | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 4 | 3
Sepsis (Infections and infestations) | 3 | 2
Bacteraemia (Infections and infestations) | 1 | 3
Pneumonia (Infections and infestations) | 2 | 1
Urinary Track Infection (Infections and infestations) | 1 | 2
Gastroenteritis Viral (Infections and infestations) | 1 | 1
Septic Shock (Infections and infestations) | 0 | 2
Catheter Related Infection (Infections and infestations) | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Escherichia Bacteraemia (Infections and infestations) | 0 | 1
Klebsiella Infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 0 | 1
Viral Oesophagitis (Infections and infestations) | 0 | 1
Mucosal Inflammation (General disorders) | 0 | 6
Chest Pain (General disorders) | 2 | 2
Pyrexia (General disorders) | 4 | 0
Asthenia (General disorders) | 1 | 2
Catheter Thrombosis (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Multi-Organ Failure (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Venous Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 5 | 2
Hypertension (Vascular disorders) | 1 | 2
Hypertensive Crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Jugular Vein Thrombosis (Vascular disorders) | 1 | 0
Vena Cava Thrombosis (Vascular disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 2
Bundle Branch Block Left (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Tamponade (Cardiac disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 4 | 2
Acute Prerenal Failure (Renal and urinary disorders) | 0 | 1
Calculus Ureteric (Renal and urinary disorders) | 1 | 0
Ureteric Obstruction (Renal and urinary disorders) | 1 | 0
Anastomotic Complication (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional Hernia (Injury, poisoning and procedural complications) | 1 | 0
Wound Complication (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour Local Invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Conversion Disorder (Psychiatric disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 0 | 1
Violence-Related Symptom (Psychiatric disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Hepatic Encephalopathy (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | XELOX Q3W + Bevacizumab (N=208) | XELOX Q2W + Bevacizumab (N=211)
Diarrhoea (Gastrointestinal disorders) | 131 | 152
Nausea (Gastrointestinal disorders) | 117 | 139
Vomiting (Gastrointestinal disorders) | 74 | 81
Abdominal Pain (Gastrointestinal disorders) | 55 | 49
Constipation (Gastrointestinal disorders) | 36 | 39
Dyspepsia (Gastrointestinal disorders) | 16 | 25
Stomatitis (Gastrointestinal disorders) | 16 | 24
Abdominal Pain Upper (Gastrointestinal disorders) | 13 | 12
Flatulence (Gastrointestinal disorders) | 12 | 10
Fatigue (General disorders) | 123 | 105
Temperature Intolerance (General disorders) | 37 | 34
Mucosal Inflammation (General disorders) | 15 | 32
Pyrexia (General disorders) | 22 | 25
Asthenia (General disorders) | 14 | 16
Oedema Peripheral (General disorders) | 11 | 13
Neuropathy Peripheral (Nervous system disorders) | 67 | 57
Peripheral Sensory Neuropathy (Nervous system disorders) | 51 | 40
Headache (Nervous system disorders) | 31 | 27
Paraesthesia (Nervous system disorders) | 27 | 25
Dizziness (Nervous system disorders) | 20 | 16
Dysgeusia (Nervous system disorders) | 15 | 18
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 50 | 86
Rash (Skin and subcutaneous tissue disorders) | 21 | 25
Dry Skin (Skin and subcutaneous tissue disorders) | 26 | 15
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 8 | 13
Skin Reaction (Skin and subcutaneous tissue disorders) | 6 | 14
Anorexia (Metabolism and nutrition disorders) | 51 | 58
Dehydration (Metabolism and nutrition disorders) | 28 | 34
Hypokalaemia (Metabolism and nutrition disorders) | 33 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 24
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 23
Hiccups (Respiratory, thoracic and mediastinal disorders) | 11 | 10
Anaemia (Blood and lymphatic system disorders) | 36 | 22
Neutropenia (Blood and lymphatic system disorders) | 21 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 26 | 9
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 23 | 18
Back Pain (Musculoskeletal and connective tissue disorders) | 14 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 6
Insomnia (Psychiatric disorders) | 25 | 24
Anxiety (Psychiatric disorders) | 10 | 18
Depression (Psychiatric disorders) | 11 | 17
Weight Decreased (Investigations) | 31 | 45
Urinary Tract Infection (Infections and infestations) | 11 | 13
Upper Respiratory Tract Infection (Infections and infestations) | 10 | 11
Hypertension (Vascular disorders) | 23 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.